CLINICAL TRIAL: NCT00458627
Title: Body Plethysmograph Measurements Before and After Methacholine Challenge in Early Childhood
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: 2044-CTIL
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Asthma
Keywords: Plethysmograpy; preschool; methacholine challenge; spirometry; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In our previous study of Methacholine Challenge Tests (MCT) in preschool children, we found that wheeze detection was associated with significant reduction in flows and vital capacity values. We hypothesized that this finding is associated with trapped-air rather than the children's loss of cooperation/concentration.

Objectives: To test this hypothesis by attempting plethysmography measurements during MCT.

DETAILED DESCRIPTION:
In young children that cannot perform adequately spirometry methacholine challenge test (MCT) is continued until any of the following clinical signals occurred: appearance of audible wheeze, a fall of >5% in O2-saturation, or an increase of >50% in respiratory rate and/or heart rate. In our previous study [1] we assessed the feasibility of determining PC20-FEV1 in relation to audible wheeze detection during MCT in asthmatic preschool children. We found that at end of test (EOT), the reduction in flows of the forced expiratory flow volume (FEFV) curves was accompanied by reduction in forced vital capacity (FVC) though reductions in flows were higher than the reduction in volume. We hypothesized that this finding is associated with trapped-air rather than the children's loss of cooperation or concentration. We have also thought that determining lung volume by whole body plethysmograpy, has the advantage of measuring airway resistance in relation to FRC. Hence, plethysmographic measurements of lung volumes during MCT may shed light on the physiological relation between airway obstruction and hyperinflation at the end of MCT when audible wheeze is detected. However, plethysmography requires the patient's cooperation and coordination to perform brief panting maneuvers against closed airways. So far, only airway resistance has been measured in the plethysmograph [10], as it is believed that young children will not comply with the occlusions needed for lung volume measurements within the plethysmograph.

The aims of the present study were twofold: a) to test if young children are capable of performing plethysmographic maneuvers required for FRC measurements; and b) to investigate if the reduction in vital capacity at maximal reduction in flows of the FEFV curves, found at wheeze detection during MCT, is due to true elevation of FRC and air trapping, or is artificially related to patients' loss of motivation/cooperation.

Methods:

Lung volumes and airway resistance will be measured in a commercial, whole body ZAN500 constant volume body plethysmograph (ZAN-Messgeraete GmbH, Germany). The plethysmograph is equipped with a graphic display for preschool children to increase cooperation. The chair can be adjusted so that the child can comfortably sit up straight with a nose-clip, and reach the mouthpiece without flexing the neck.

The plethysmography procedure will be performed according to recommendations. The test events will be explained to the child in detail outside of the plethysmograph. After that, the measurements will be carried out in the same sequence that was explained to the child. FRC will be measured by allowing for 2-3 breathing attempt series of superimposed straight lines (separated only by thermal drift). The best test out of two technically accepted series was analyzed.

MCT will be performed according to the ATS guidelines for the Methacholine Challenge Test. Tests will be performed in a designated room at the Pediatric Pulmonary Unit, Meyer Children's Hospital, Haifa, Israel. A parent and the investigating team will be present throughout the test. Tests will be performed with triple doses of fresh Methacholine solutions (0.057 to13.395 mg/ml) dissolved in saline. Solutions will be driven by a KoKo-PDS dosimeter (Ferraris Respiratory, Louisville, CO) via mouthpiece while the child was sitting upright with a nose-clip and breathing at least 10 deep breaths. Five-minute intervals will be taken between concentrations until the maximal concentration or the end point will be reached (see below). Oxygen saturation and heart-rate will be monitored continuously by pulse-oximetry (Ohmeda Biox 3700 Pulse Oximeter, USA). Auscultation for 20-seconds over the trachea and two zones of both lungs (upper front and lower back) will be performed according to recommendation. The following indices will be considered as EOT: appearance of audible wheeze, a fall of 5% in O2-saturation, or an increase of 50% in respiratory rate and/or heart rate. Nebulized Albuterol (2.5mg) was administrated after lung function measurements.

Spirometry: FEFV curves will be measured with a KoKo PDS commercial spirometer (Ferraris Respiratory, Louisville, CO), using the program incentives targets (peak expiratory flow rates or vital capacity). Calibration was performed before the testing sessions. The curves will be monitored on the computer screen to ensure best effort. On-line rejection of curves will be based on published quality control for older and preschool children including visual inspection for "non-cooperation" errors, which included poor effort, incomplete expiration, cough and glottis closure. Acceptable curves had to show a rapid rise to peak flow, and a gradual, smooth decline of flow down to residual volume.

Sequence of lung function tests: Baseline measurements included spirometry followed by plethysmography. After baseline measurements MCT will be performed. A duplicate spirometry set will be performed immediately after auscultation and during the interval between inhalations. Plethysmography will be repeated following the last spirometry at EOT and after auscultation.

ELIGIBILITY:
Inclusion Criteria:

* 2.5-6.9 year-old children who were asthmatic according to GINA guidelines.
* All children previously had recurrent episodes of wheeze, cough and/or shortness of breath with clinical response to bronchodilator.
* Children were included only if they had not received anti-inflammatory medication for at least one week prior to the test or bronchodilators for at least 24 hours prior to the study.
* On the day of testing, children were included if they had normal chest auscultation and FEV1>75% predicted for healthy preschool children.

Exclusion Criteria:

* Presence of other chronic respiratory conditions
* Emergency room visit in the past three months
* Respiratory infection in the past month

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2006-02; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Rambam medical Center, Haifa, Israel; Daphna Vilozni, PhD, Principal Investigator — Rambam Health Care Campus

REFERENCES:
- [Background] Bentur L, Beck R, Elias N, Barak A, Efrati O, Yahav Y, Vilozni D. Methacholine bronchial provocation measured by spirometry versus wheeze detection in preschool children. BMC Pediatr. 2005 Jun 28;5:19. doi: 10.1186/1471-2431-5-19. PMID 15985169
- [Background] Vilozni D, Barak A, Efrati O, Augarten A, Springer C, Yahav Y, Bentur L. The role of computer games in measuring spirometry in healthy and "asthmatic" preschool children. Chest. 2005 Sep;128(3):1146-55. doi: 10.1378/chest.128.3.1146. PMID 16162700
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836